CLINICAL TRIAL: NCT03455348
Title: Impact of Radial Arterial Location on Arterial Catheter Lifetime in Surgical Intensive Care
Acronym: KARTDISCHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KARTDISCHO
Record Dates: First submitted 2017-10-04; First posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2017-12

CONDITIONS: Dysfunctions Arterial Catheter
MeSH Terms: interventions — Catheterization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cathete to less than 4 four centimeters to the wrist joint (No Intervention)
- catheter to more than four centimeters to the wrist joint (Active Comparator)
  Interventions: Other: catheter insertion

INTERVENTIONS:
Other: catheter insertion — catheter insertion one to less than 4 four centimeters to the wrist joint (Group A) and the other, to more than four centimeters to the wrist joint. (Group B)
  Arms: catheter to more than four centimeters to the wrist joint

SUMMARY:
Dysfunctions radial arterial catheter are frequent. This was a prospective, randomized observational study monocentric in ICU in France. Patients are randomized in 2 groups : One to less than 4 four centimeters to the wrist joint (Group A) and the other, to more than four centimeters to the wrist joint. (Group B). The primary outcome was the incidence of catheter dysfunction (defined by the impossibility of taking blood from the catheter and / or the impossibility having a reliable blood pressure curve). Investigators compared also the incidence of infection, satisfaction of doctors and nurses, the numbers of days with catheter and the cause of withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted in ICU, older than 18 years and who required an arterial catheter are include

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
the incidence of dysfunction motivating catheter removal as a function of the distance from the carpal radio joint. | through study completion- 2 months
  The dysfunction is defined by the impossibility of taking blood from the catheter and / or the impossibility having a reliable blood pressure curve